CLINICAL TRIAL: NCT01875393
Title: Study of the Efficacy,Safety and Quality of Life After TOOKAD® Soluble Vascular Targeted Photodynamic Therapy (VTP) for Minimally Invasive Treatment of Localized Prostate Cancer
Brief Title: Efficacy,Safety and Quality of Life After TOOKAD® Soluble VTP for Localized Prostate Cancer
Acronym: PCM304
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1201 PCM304
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Prostatic Disease; Genital Neoplasm,male; Urogenital neoplasm; Genital disease,male; Male urogenital disease; Neoplasms; Neoplasms by site; Prostatic neoplasm; Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Carcinoma | interventions — padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TOOKAD® Soluble (Experimental): TOOKAD® Soluble, lyophilized formulation,given at a dose of 4 mg/kg.
  Interventions: Drug: TOOKAD® Soluble

INTERVENTIONS:
Drug: TOOKAD® Soluble — The VTP procedure will consist of a single, 10 minute infusion of 4mg/kg TOOKAD® Soluble. The drug will be activated by laser light at 753nm, with a fixed energy of 200Joules/cm, and a fixed power of 150mWatts/cm, delivered through transperineal interstitial optical fibers. The needles are positioned in the prostate under ultra sound image guidance.
  Other Names: WST11

SUMMARY:
The aim of this study is to confirm the Efficacy,the Safety and the Quality of Life after TOOKAD® Soluble VTP in localized prostate cancer patients.

DETAILED DESCRIPTION:
The study is designed as a multicenter, single-arm, open label, 12 months follow-up clinical trial. Men with localized prostate cancer will be treated with TOOKAD® Soluble VTP under general anesthesia.

Patients will be followed-up for 12 months with patient questionnaires on QoL, erectile and urinary functions, clinical evaluation with study visits at 1, 3, 6 and 12 months , Prostate Specific Antigen(PSA) testing at 3, 6 and 12 months. In addition, they will have biopsy at 6 months (± 2) and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven localized prostate carcinoma diagnosed using prostate biopsy showing:

  * Gleason 3+3 prostate
  * Gleason 3+4 prostate adenocarcinoma is acceptable provided it is not present in more than 2 cores and no more than 50% cancer in any core.
* Clinical stage up to cT2a - N0/Nx - M0/Mx.
* Serum prostate-specific antigen (PSA) ˂ 20ng/ml
* Prostate volume ≥ 25 cc and ≤ 70 cc.
* Male subjects aged 18 years or older.
* Signed Informed Consent Form by the patient.

Exclusion Criteria:

* Unwillingness to accept the treatment.
* Any prior or current treatment for prostate cancer, including surgery, radiation therapy (external or brachytherapy)or chemotherapy.
* Any surgical intervention for benign prostatic hypertrophy.
* Any condition or history of illness or surgery that may pose an additional risk to men undergoing the VTP procedure.
* Life expectancy less than 10 years.
* Participation in another clinical study involving an investigational product within 1 month before study entry.
* Subject unable to understand the patient's informed consent document, to give consent voluntarily or to complete the study tasks, especially unable to understand and fulfill the health-related QoL questionnaire.
* Subject in custody and or in residence in a nursing home or rehabilitation facility.
* Any condition or history of active rectal inflammatory bowel disease or other factors which may increase the risk of fistula formation;
* Any hormonal manipulation (excluding 5-alpha-reductase inhibitors) that alters androgen production or use of androgen supplements within the previous 6 months;
* Any history of urethral stricture disease;
* Any history of acute urinary retention within 6 months of study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To confirm that a significant proportion of patients will be prostate cancer free on the biopsy. | Month 12
  Number of patients with a negative biopsy.

SECONDARY OUTCOMES:
Changes in urinary and erectile functions and their potential impact on quality of life using International Prostate Symptom Score (IPSS), International Index of Erectile Function (IIEF) and the General quality of life (EQ5D) questionnaires. | Screening, 1, 3, 6 and 12 months after completing treatment
  Patients' reported outcome measures (PROMs) impairment: urinary symptoms using IPSS and erectile functions using IIEF. Quality of life using EQ5D will also be described
The rate of adverse events. | Screening-Month 12
  Adverse event reporting.
The overall cancer burden in the prostate determined by biopsy as compared to baseline. | Month 12
  Total length of cancer present in all cores taken in any given biopsy session
The rate of severe prostate cancer related events: cancer extension to T3, metastasis and prostate cancer related death | Screening-Month 12
  Severe prostate cancer related events: cancer extension to T3, metastasis or prostate cancer-related death.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Arturo Rodriguez Rivera, Dr, Principal Investigator — Hospital General Tlahuac; Mary Lol Ve Mendoza Medina, Dr, Principal Investigator — Hospital General Tlahuac; Luis Zegarra Montes, Professor, Principal Investigator — Hospital Nacional Cayetano Heredia; Ramón Rodriguez, Professor, Principal Investigator — Pan-American Medical Research Institute (PAMRI) then moved to Consultario del Dr Rodriguez
Locations (3):
- Hospital General Tlahuac, Mexico City, Mexico
- Pan-American Medical Research Institute (PAMRI) then moved to Consultario del Dr Rodriguez, Panama City, Panama
- Hospital Nacional Cayetano Heredia, San Martín de Porres, Peru

IPD SHARING:
Plan to Share IPD: Yes
The data are available in case report form for each patient

REFERENCES:
- [Derived] Azzouzi AR, Barret E, Bennet J, Moore C, Taneja S, Muir G, Villers A, Coleman J, Allen C, Scherz A, Emberton M. TOOKAD(R) Soluble focal therapy: pooled analysis of three phase II studies assessing the minimally invasive ablation of localized prostate cancer. World J Urol. 2015 Jul;33(7):945-53. doi: 10.1007/s00345-015-1505-8. Epub 2015 Feb 25. PMID 25712310